CLINICAL TRIAL: NCT07383584
Title: Sleep Banking Pre-Surgery for Improved Chronic Post-Surgical Pain: A Pilot Study
Brief Title: The Impact of Extending Sleep Before Joint-replacement Surgery on Post-surgical Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USUHS 2025-158
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Joint (Knee or Hip Replacement)
Keywords: sleep banking; sleep extension; chronic pain; recovery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Sleep banking compared to sleep as usual (no intervention)
Who Masked: Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep extension (Experimental): The sleep extension group will add 2 h of sleep per night the week before surgery
  Interventions: Behavioral: Sleep banking
- Habitual sleep (No Intervention): The habitual sleep group maintain their usual hours of sleep per night the week before surgery

INTERVENTIONS:
Behavioral: Sleep banking — The sleep extension group will add 2 hour of sleep per night the week before surgery
  Arms: Sleep extension

SUMMARY:
This study will evaluate the impact of sleep banking on joint replacement surgery recovery.

DETAILED DESCRIPTION:
Sleep is emerging as a target for pain management. The purpose of this study is to determine the feasibility and efficacy of extending sleep (sleep "banking") on self-reported pain outcomes post-surgery. This is a prospective, interventional, between-subjects, randomized study with a control condition. Participants will be patients undergoing knee or hip replacement surgery at Naval Medical Center San Diego. Participants will be randomized to either a sleep banking group, where they attempt to extend nightly sleep in the week leading up to surgery, or to a habitual sleep control group, sleeping in their typical pattern for that same period. Sleep and pain will be monitored daily yn the two weeks pre- and one week post-surgery. After that, they will be sent electronic follow-up sleep and pain questionnaires at 1, 3, 6, 9, and 12 weeks post-surgery. Participants in the sleep banking group will also complete additional questionnaire items on the feasibility and implementation of the sleep banking protocol. Feasibility of sleep banking will be assessed by examination of the sleep between groups during the intervention week, as well as by the analysis of the implementation questions. Efficacy will be assessed by examination of self-reported pain outcomes post-surgery by group. The primary hypothesis is that self-reported pain outcomes will be improved in the sleep banking group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals scheduled for a joint replacement surgery (knee or hip) at Naval Medical Center San Diego
* Aged 18-74 years

Exclusion Criteria:

* Individuals < 18 or >74 years of age at enrollment
* Individuals diagnosed with untreated sleep disorders
* Individuals with scheduled timezone travel or work schedule changes (>/= 3 hour time change) in the two weeks before surgery

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Weeks 1-15
  Defense and Veterans Pain Rating Scale. On a scale of 0-10, with higher scores denoting more pain.
Pain Medication Use | Weeks 1-15
  Opioid Use Diary

SECONDARY OUTCOMES:
Physical Function | Weeks 1-15
  Patient-Reported Outcomes Measurement Information System (PROMIS) -29 Adult Profile 2.0 Instrument, Physical Function subscale. Each item is scored on a scale 1-5, with 1=without any difficulty and 5=unable to do. Items will be summed and t-scored (0-100), with higher scores denoting less function.
Sleep Disturbance | Weeks 1-15
  Patient-Reported Outcomes Measurement Information System (PROMIS) -29 Adult Profile 2.0 Instrument, Sleep Disturbance subscale. Each item is scored on a scale 1-5, with 1=not at all and 5=very much. Items will be summed and t-scored (0-100), with higher scores denoting more sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No